CLINICAL TRIAL: NCT04744649
Title: Efficacy and Safety of Neoadjuvant Immunotherapy and Chemotherapy for Locally Advanced Esophagogastric Junction and Gastric Cancer : a Open-label, Phase 2 Randomised Controlled Trial (NICE Trial)
Brief Title: Neoadjuvant Immunotherapy and Chemotherapy for Locally Advanced Esophagogastric Junction and Gastric Cancer Trial
Acronym: NICE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Guoxin Li, President, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NICE
Record Dates: First submitted 2021-01-23; First posted 2021-02-09 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Gastric Cancer; Stomach Neoplasm
Keywords: Gastric Cancer; Esophagogastric Junction Cancer; Immunotherapy and Chemotherapy; Neoadjuvant
MeSH Terms: conditions — Stomach Neoplasms | interventions — XELOX; Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): The patients with combined positive score (CPS) of PD-L1 protein expression≥5 were randomised to control group(N=40), will receive the neoadjuvant regime of XELOX or SOX.
  XELOX: Oxaliplatin+Capecitabine; SOX: Oxaliplatin+S-1. Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3w; S-1:40~60mg Bid, d1~14, q3w; Capecitabine: 1000mg/m2 Bid, d1-14, q3w; Neoadjuvant chemotherapy for 4 cycles, adjuvant chemotherapy for 4 cycles.
  Interventions: Drug: XELOX or SOX
- Experimental group (Experimental): The patients with combined positive score (CPS) of PD-L1 protein expression≥5 were randomised to experimental group(N=40), will receive the neoadjuvant regime of JS001+XELOX or SOX.
  XELOX: Oxaliplatin+Capecitabine; SOX: Oxaliplatin+S-1. JS001: 240mg, ivdrip, d1, q3w; S-1:40~60mg Bid, d1~14, q3w; Capecitabine: 1000mg/m2 Bid, d1-14, q3w; Neoadjuvant chemotherapy for 4 cycles, adjuvant chemotherapy for 4 cycles.
  Interventions: Drug: JS001+XELOX or SOX
- Exploratory group (Other): All the patients of Epstein-Barr virus-positive (EBV(+)) [N=15]or mismatch repair-deficient (dMMR)/ microsatellite instability-high (MSI-H)[N=15] , will be assigned to exploratory group, and will receive the neoadjuvant regime of JS001+XELOX or SOX.
  XELOX: Oxaliplatin+Capecitabine; SOX: Oxaliplatin+S-1. JS001: 240mg, ivdrip, d1, q3w; S-1:40~60mg Bid, d1~14, q3w; Capecitabine: 1000mg/m2 Bid, d1-14, q3w; Neoadjuvant chemotherapy for 4 cycles, adjuvant chemotherapy for 4 cycles.
  Interventions: Drug: JS001+XELOX or SOX

INTERVENTIONS:
Drug: XELOX or SOX — XELOX: Oxaliplatin+Capecitabine; SOX: Oxaliplatin+S-1
  Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3w;
  S-1:40~60mg Bid, d1~14, q3w;
  Capecitabine: 1000mg/m2 Bid, d1-14, q3w;
  Neoadjuvant chemotherapy for 4 cycles, adjuvant chemotherapy for 4 cycles.
  Drug: Oxaliplatin Oxaliplatin: 130mg/m2，iv drip for 2h，d1, q3w
  Drug: S1 S-1: 40~60mg Bid，d1~14, q3w
  Drug: Capecitabine Capecitabine: 1000mg/m2 Bid, d1-14, q3w Other Name: XELODA
  JS001: 240mg, ivdrip, d1, q3w;
  S-1:40~60mg Bid, d1~14, q3w;
  Capecitabine: 1000mg/m2 Bid, d1-14, q3w;
  Neoadjuvant chemotherapy for 4 cycles, adjuvant chemotherapy for 4 cycles.
  Drug: JS001 JS001, recombinant humanized anti-PD-1 monoclonal antibody for injection; 240mg ivdrip, d1, q3w.
  Other Name: PD-1 antibody
  Drug: Oxaliplatin Oxaliplatin: 130mg/m2,iv drip for 2h, d1, q3w
  Drug: S1 S-1: 40~60mg Bid,d1~14, q3w
  Drug: Capecitabine Capecitabine: 1000mg/m2 Bid, d1-14, q3w Other Name: XELODA
  Other Names: Control group
  Arms: Control group
Drug: JS001+XELOX or SOX — XELOX: Oxaliplatin+Capecitabine; SOX: Oxaliplatin+S-1
  JS001: 240mg, ivdrip, d1, q3w;
  S-1:40~60mg Bid, d1~14, q3w;
  Capecitabine: 1000mg/m2 Bid, d1-14, q3w;
  Neoadjuvant chemotherapy for 4 cycles, adjuvant chemotherapy for 4 cycles.
  Drug: JS001 JS001, recombinant humanized anti-PD-1 monoclonal antibody for injection; 240mg ivdrip, d1, q3w.
  Other Name: PD-1 antibody
  Drug: Oxaliplatin Oxaliplatin: 130mg/m2,iv drip for 2h, d1, q3w
  Drug: S1 S-1: 40~60mg Bid,d1~14, q3w
  Drug: Capecitabine Capecitabine: 1000mg/m2 Bid, d1-14, q3w Other Name: XELODA
  Other Names: Experimental group and Exploratory group
  Arms: Experimental group; Exploratory group

SUMMARY:
For locally advanced esophagogastric junction and gastric cancer (cT3-4aNxM0 or cT2N+M0), neoadjuvant chemotherapy can downstage T and N stage,treated distant micrometastases early before local therapy has begun, and finally improve the long-term survival. Combination of perioperative PD-1 antibody and chemotherapy for locally advanced esophagogastric junction and gastric cancer could be a novel therapy to increase response rate and reduce recurrence rate. JS001 in this study is a Chinese anti-PD-1 monoclonal antibody for injection which has been approved for melanoma. This study is a multi-center, open-label, randomized phase II clinical trial to evaluate safety and efficacy of JS001 in combination with perioperative chemotherapy in locally advanced esophagogastric junction and gastric cancer. Differences in gut microbiome and tumor immune microenvironment were detected to screen people who were more sensitive to immunotherapy.

DETAILED DESCRIPTION:
Gastric cancer (GC) is one of the leading causes of cancer-related deaths worldwide and a substantial global health burden. Surgery is the only possible way to cure gastric cancer, however, more than 80% of the Chinese patients are diagnosed at advanced stages. Locally advanced esophagogastric junction and gastric cancer (cT3-4aNxM0 or cT2N+M0) could be cured by multi-disciplinary therapies including surgery, chemotherapy and radiotherapy. Neoadjuvant chemotherapy can downstage T and N stage, treated distant micrometastases early before local therapy has begun, and finally improve the long-term survival. However, the therapeutic effects remain unsatisfactory. PD-1 antibody has demonstrated its efficacy in metastatic gastric cancer and has been proved to be effective in neoadjuvant setting in lung cancer and melanoma. Combination of perioperative PD-1 antibody and chemotherapy for locally advanced esophagogastric junction and gastric cancer could be a novel therapy to increase response rate and reduce recurrence rate. JS001 in this study is a Chinese anti-PD-1 monoclonal antibody for injection which has been approved for melanoma. This study is a multi-center, open-label, randomized phase II clinical trial to evaluate safety and efficacy of JS001 in combination with perioperative chemotherapy in locally advanced esophagogastric junction and gastric cancer. Differences in gut microbiome and tumor immune microenvironment were detected to screen people who were more sensitive to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed) informed consent;
2. Age ≥ 18 years and ≤75 years.
3. Confirmed gastric and gastroesophageal junction adenocarcinoma by Gastroscopic biopsy histopathological examination.
4. Imaging (CT/MRI) and diagnostic laparoscopy confirmed at the stage of cT3/4a Nx or T2 N+, M0(AJCC 8th) before randomization.
5. confirmed by immunohistochemistry (IHC) staining or genetic and transcriptional profiling detection to meet one of the following conditions:

   1. Combined positive score (CPS) of PD-L1 protein expression ≥5.
   2. Epstein-Barr virus-positive (EBV(+)).
   3. mismatch repair-deficient (dMMR).
   4. Microsatellite instability-high (MSI-H)
6. The Eastern Cooperative Oncology Group Performance status (ECOG PS) 0-1
7. Expected survival period ≥ 12 weeks
8. The main organ function meets the following criteria within 7 days before treatment:

   1. Hemoglobin (Hb) level ≥9.0 g/dl
   2. Neutrophil count (ANC)≥1.5×l09/L
   3. Platelet (PLT) ≥100×109/L
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN
   5. Alkaline phosphatase(ALP)level ≤2.5×ULN
   6. Serum creatinine (Cr) level ≤1.5×ULN and creatinine clearance ≥60 ml/min
   7. Thyroid stimulating hormone (TSH) level ≤1×ULN (if abnormal, should require normal serum free thyroid hormone (T4) and Normal serum free triiodothyronine (T3))

Exclusion Criteria:

1. Confirmed at stage IV (AJCC 8th) or unresectable by investigator before randomization.
2. Prior chemotherapy, radiotherapy, surgery immunotherapy or molecular targeted therapy for gastric cancer;
3. Patients who have HER2 positive confiemed with IHC3+ or IHC2+ and FISH positive
4. Patients are allergic to study medication and its ingredients
5. Patients with a history of following treatments:

   1. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent
   2. Prior therapy with tyrosine kinase inhibitor within 2 weeks.
   3. Patients who have participated in other clinical trials of anti-tumor drugs within four weeks
   4. Have vaccination with attenuated live vaccines within 4 weeks prior to initiation of the study treatment or plan to vaccinate during the study;
   5. Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalent for replacement therapy
6. Patients have experienced or currently has other malignancies within 5 years.
7. Patients have an active or history of autoimmune disease that may recur or require immunosuppressive drugs within 2 weeks or less or during the study. Or have a history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation
8. Patients with other severe acute or chronic conditions that may increase the risk of participation in the study and study treatment, or may interfere with interpretation of study results, and judged by the investigator as not suitable for participation in this clinical trial.
9. Within 2 weeks or 2 weeks before randomization, patients have an active or uncontrollable infection that requires systemic antibiotic treatment
10. Diagnosed with interstitial pneumonia, non-infectious pneumonia, pulmonary fibrosis, acute lung disease;
11. Patients with active tuberculosis or receiving previous anti-tuberculosis therapy within one year
12. Women who are pregnant, breast-feeding or planning to become pregnant during treatment or within 6 months after treatment ends.
13. Patients have a history of psychotropic substance abuse and are unable to quit or have a mental disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 14 weeks
  It is defined as residual tumors less than 10% after neoadjuvant immunotherapy and(or) chemotherapy

SECONDARY OUTCOMES:
Disease-free survival (DFS) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  The Kaplan-Meier survival from the initiation date of first cycle until the date of first documented recurrence.
Overall survival(OS) | From date of randomization until the date of first documented date of death from any cause, assessed up to 36 months
pCR | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 14 weeks
  Pathological complete response after neoadjuvant immunotherapy and(or) chemotherapy
R0 resection rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 14 weeks
  Rate of microscopically margin-negative resection
Adverse event incidence rate | Patients will be assessed for adverse events throughout the study at every visit during treatment and at 3-month follow-up visit (3 months after treatment ends)
  Number of participants with treatment-related adverse events as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D., Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University; Liying Zhao, M.D., Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (10):
- China (10):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The six affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, the Second Affiliated Hospital of Guangzhou University of Chinese Medicine,, Guangzhou, Guangdong
  - Mao ming people's hospital, Maoming, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Eighth Affiliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: Yes
We will share Study Protocol and Statistical Analysis Plan (SAP)
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Zhao L, Liu H, Yu J, Yuan S, Liang H, Wang W, Jiang J, Yu L, Liang L, Chen Z, Chen X, Zhong X, Zheng Y, Li F, Lin T, Zhao M, Chen T, Chen H, Hu Y, Li G. Efficacy and safety of neoadjuvant toripalimab plus chemotherapy in localized deficient mismatch repair/microsatellite instability-high gastric or esophagogastric junction adenocarcinoma (NICE): a multicentre, single-arm, exploratory phase 2 study. EClinicalMedicine. 2025 Aug 12;87:103421. doi: 10.1016/j.eclinm.2025.103421. eCollection 2025 Sep. PMID 40838201